CLINICAL TRIAL: NCT04207125
Title: Improving ImmunoSuppression Adherence After Liver or Kidney Transplantation -a Randomized Controlled Single Centre Trial
Brief Title: Improving ImmunoSuppression Adherence After Liver or Kidney Transplantation
Acronym: ISALK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32-062 ex 19/20
Record Dates: First submitted 2019-11-20; First posted 2019-12-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Adherence Intervention Post Transplantation
MeSH Terms: interventions — Sex Education

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without multilevel intervention (No Intervention): patients after liver or kidney transplantation / standard care
- With multilevel intervention (Active Comparator): patients after liver or kidney transplantation / multilevel intervention program
  Interventions: Behavioral: Multilevel psychotherapeutic intervention programme

INTERVENTIONS:
Behavioral: Multilevel psychotherapeutic intervention programme — Part 1: Educational Training and Mentoring After transferring the patient from the intensive care unit to the transplant surgery unit, nurses are planning a nursing diagnosis called "therapy recommendations and coping strategies, effective implementation". 3 days after the transfer, nurses start to give information twice a day (morning and evening) about the medication, which the patients are currently taking. The nurse is also handing out a folder, which contains information about the multilevel intervention programme.
  Individual Treatment Approach Patients, who seem to be non-adherent during their outpatient follow-ups, are contacted through the co-investigators for a one-to-one session. The content of this session is to promote patients engagement in self-management of their chronic illness. The goal of the treatment is to improve the individual's ability to manage symptoms, treatments, physical and psychosocial consequences and lifestyle changes.
  Other Names: education training
  Arms: With multilevel intervention

SUMMARY:
Indication: liver (LT) or kidney Transplantation (KT)

Objectives: to measure medication adherence in liver or kidney transplant patients with and without multilevel intervention programme over time

Trial Design: prospective, single-centre, randomized controlled study

Population: patients (male/female/diverse) between 18 and 90 years of age scheduled for LT or KT

Sample Size:

75 control patients (standard of care) 75 patients in treatment group (participation in multilevel intervention programme)

Statistical Analysis: The data will be analysed descriptively; continuous variables will be summarized using mean ± SD (standard deviation) or median, minimum and maximum and categorical data will be summarized using absolute and relative frequencies. For the primary outcome (Adherence to the immunosuppressive regime measured by BAASIS) and further categorical variables, differences between the groups will be assessed by the Pearson Chi-square test or Fisher's exact test. Group differences for continuous parameters will be assessed by the two-sample T-test or Mann-Whitney-U-test as appropriate.

Trial Duration and Dates: November 2019-October 2021

DETAILED DESCRIPTION:
Organ transplantation is the best option for patients with chronic organ failure. After kidney (KT) or liver transplantations (LT), immunosuppressive medications have to be taken to avoid rejection. Lifelong adherence, the extent to which the patients behaviour matches the agreed upon prescribers recommendations, to immunosuppressive drugs is important to prevent graft failure (Pabst et al., 2015). The consequent immunosuppression intake and regular physician visits are important factors for a long transplant survival (Nöhre et al., 2018).

A high rate of immunosuppressive medication non-adherence and its impact on post-transplant graft function indicate a need for adherence enhancing interventions (De Bleser et al., 2011).

Non-adherence is linked to poor post-transplant outcomes including late acute rejection and graft loss (De Geest S. et al 2011; Dew MA et al 2008). Dew et al. concluded from a meta- analysis of 147 transplantation studies that nonadherence in renal allograft recipients was highest among solid organ transplant recipients, reaching 36 cases per 100 patients per year (Dew et al., 2007). Detection of adherence can be obtained by objective direct measures (observation that medication was taken) or indirect and subjective measures like self-reporting. The indirect measures include serum drug levels, biological markers and electronic monitoring. Adherence is a dynamic process with the need to be repetitive over time. The monitoring should be incorporated into the routine clinical management of all organ recipients. A recent study showed that combining self-reporting, assay and clinicians report yielded the highest sensitivity (72%) and specificity (42%) when compared to electronic monitoring (Low et al., 2019). Some new evidence suggest that moving from twice-daily to once-daily dosing of the immunosuppressive regimen, the calcineurin inhibitor, show indifferent prevalence rates with increased adherence or not improving the adherence (Lehner et al., 2018; Fellström et al., 2018).The aim of our study is to test the efficacy of such a multilevel education and psychosomatic intervention programme for improving medication adherence in patients after LT or KT.

1. Primary Objective and Primary Endpoint The primary endpoint is the assessment of patient adherence using a validated version of the Basel Assessment of Adherence to Immunosuppressive Medication Scale (BAASIS) questionnaire.
2. Secondary Objectives and Secondary Endpoints Secondary endpoints include the influence of the multilevel intervention programme on the coefficient of variation (CV%) of Tacrolimus (TAC), clinical outcomes including incidence of infections, acute rejection, liver and kidney values, death, graft loss, hospital readmission during the study period, side effects, number of trough level controls necessary during first 6 months, and achievement of TAC target concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male/female) listed for LT and KT
* Ability of subject to understand character and individual consequences of the trial
* Fluent in speaking the German language
* Written informed consent must be available before enrolment in the trial
* Basis immunosuppression with Tacrolimus

Exclusion Criteria:

* Patients < 18 or > 90 years
* Pregnant or lactating women
* Refusal to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-09-07 (Estimated); Study Completion 2021-09-07 (Estimated)

PRIMARY OUTCOMES:
self-rating of adherence | 6 months
  Basler Assessment of Adherence to Immunosuppressive Medication Scale (BAASIS) The Basler assessment was developed to assess adherence to immunosuppressive drugs in adult transplant recipients. It follows the newly published taxonomy of medication adherence. This self-reported interview consists of three quantifiable phases: initiation, implementation and persistence. Five Items assess the implementation dimension and one assesses the persistence. An optional item assesses initiation. Responses to four questions are given on a 6-point scale ranging from zero (never) to five (every day) (Dobbels et al., 2010).

SECONDARY OUTCOMES:
Coefficient of Variation (CV%) of Tacrolimus | 6 months
Occurrence of infection episodes | 6 months
Occurrence of rejection episodes | 6 months
  Biopsy-proven acute rejection
Rejection therapy | 6 months
  Administered rejection therapies
Occurrence of side effects | 6 months

OTHER OUTCOMES:
influencing psychodynamic factors | 6 months
  Survey on distress: Global Symptom Load Level of Personality Functioning The Relationship Structures questionnaire of the Experiences in Close Relationships-Revised (ECR-RS) Scale that is designed to assess attachment dimensions in multiple contexts will be used (Frayley, Heffernan, & Vicary et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schemmer, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Klin. Abteilung für Transplantationschirurgie, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagner-Skacel J, Fink N, Kahn J, Dalkner N, Jauk E, Bengesser S, Mairinger M, Schussler G, Pieh C, Stadlbauer V, Kirsch AH, Zitta S, Rosenkranz AR, Fickert P, Schemmer P. Improving adherence to immunosuppression after liver or kidney transplantation in individuals with impairments in personality functioning - A randomized controlled single center feasibility study. Front Psychol. 2023 Mar 9;14:1150548. doi: 10.3389/fpsyg.2023.1150548. eCollection 2023. PMID 36968754